CLINICAL TRIAL: NCT03792724
Title: Phase I-II Study of Intratumoral Urelumab Combined With Nivolumab in Patients With Solid Tumors
Acronym: INTRUST
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTRUST
Record Dates: First submitted 2018-12-20; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — urelumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A (Experimental): Three doses of intratumoral urelumab will be administered, every 4 weeks. after which Nivolumab will be given at a fixed dose of 240 mg for Cycle 2 and at a fixed dose of 480 mg every 4 weeks (Q4W) from Cycle 3 and beyond
  Interventions: Drug: Urelumab + Nivolumab
- Cohort B (Experimental): Three doses of intratumoral urelumab will be administered, every 4 weeks. after which Nivolumab will be given at a fixed dose of 240 mg for Cycle 2 and at a fixed dose of 480 mg Q4W from Cycle 3 and beyond
  Interventions: Drug: Urelumab + Nivolumab

INTERVENTIONS:
Drug: Urelumab + Nivolumab — Treatment with intratumoral urelumab after which Nivolumab will be given.

SUMMARY:
Open label, phase I-II study to evaluate the safety and activity of intratumoral urelumab combined with systemic nivolumab in patients with advanced solid tumors. Serial tumor and blood samples will be obtained during the study to characterize the changes induced by treatment in the tumor microenvironment, as well as predictive biomarkers of response.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing and other requirements of the study.
3. Patients must present the following tumor types:

   1. For the phase I part, patients with any tumor type are eligible.
   2. For the phase II part, two cohorts will be established:

   i. Cohort A will include patients presenting tumor types with known sensitivity to Programmed cell death protein 1 (PD1)/ Programmed Death-ligand 1 (PDL1) blockade (e.g: melanoma, renal cancer, lung cancer, urothelial cancer, colorectal cancer presenting microsatellite instability (MSI), …). These patients must be naïve to PD1/PDL1 blockade.

   ii. cohort B will include patients with PD1/PDL1 sensitive tumors that have progressed following previous PD1/PDL1 blockade (e.g: melanoma, NSCLC, renal cancer, bladder cancer ...). Additional treatments may be administered between prior PD1/PDL1 blockade and inclusion in the study, but if administered immediately before, a minimum wash-out period of four weeks must be observed between both treatments.
4. Patients must have received standard therapy, according to investigator´s criteria, or must be ineligible for standard therapy.
5. Patients must present at least one tumor lesion that is amenable to perform sequential intratumoral therapy and biopsies.
6. Measurable disease according to RECIST criteria. The measurable lesion(s) must be different than the lesion treated with intratumoral urelumab.
7. There is no limit on previous treatment lines, as long as the other inclusion criteria are met.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
9. Life expectancy >12 weeks.
10. Adequate organ function defined by:

    1. Bone Marrow Reserve: white blood cells (WBC): >=2000/ mm3 absolute neutrophil count (ANC) >=1500x 109/L; platelet count >=100000/ mm3 100 x 109/L; hemoglobin >=9.0 g/dL).
    2. Hepatic: bilirubin <1.5 times the upper limit of normality (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3.0 x ULN (BR< 3 x ULN for patients with Gilbert´s Syndrome).
    3. Renal: creatinine <1.5 x ULN or estimated creatinine clearance > 40 ml/min, using the Cokcroft-Gault formula.
11. Women of childbearing potential (WOCBP, i.e: fertile, following menarche and until becoming post-menopausal unless permanently sterile) must use a highly effective method to avoid pregnancy (i.e: combined estrogen and progestogen associated with inhibition of ovulation (oral, intravaginal or transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable); intrauterine device; intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence for 23 weeks (30 days plus the time required for nivolumab and urelumab to undergo five half-lives) after the last dose of investigational drug.
12. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of treatment.
13. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception.
14. Patients must be at least 18 years old.

Exclusion Criteria:

1. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive the planned therapy or interfere with the interpretation of study results. Special care should be taken with conditions affecting the liver.
2. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
3. The treatment wash-out period for other previous therapies, including radiation therapy will be determined by the investigators, depending on resolution of associated toxicity. Limited-field palliative radiotherapy will not require a wash-out period. If PD1/PDL1 blockade is the previous therapy, a minimum wash-out period of four weeks must be observed between both treatments.
4. Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
5. Active brain metastasis that may interfere with interpretation of results. Subjects with controlled metastasis will be allowed to enroll. Controlled brain metastases will be defined as no radiographic progression for at least 4 weeks following radiation and/or surgical treatment.
6. Pregnant or breastfeeding patients.
7. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Routine testing is not required.
8. Positive tests for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection. Subjects with positive hepatitis C antibody and negative quantitative hepatitis C by Polymerase chain reaction (PCR) are eligible. History of resolved hepatitis A virus infection is not an exclusion criteria.
9. History of allergy to study drug components or of severe hypersensitivity reactions to any monoclonal antibodies.
10. Prisoners or subjects who are involuntarily incarcerated or who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
11. Concomitant or prior malignancy that, in the opinion of the investigator can interfere with the results of the study, in the opinion of the investigator.
12. Known drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-01-30 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | 27 months
  Number of adverse events
Recommended dose of intratumoral urelumab | 12 weeks
  mg of intratumoral urelumab
Response rate | 27 months
  Number of patients with partial response or complete response

SECONDARY OUTCOMES:
Overall survival (OS). | 27 months
  Months until death
Progression-free survival (PFS) | 27 months
  Months until progression

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Clinica Universidad de Navarra, Madrid

REFERENCES:
- [Background] Coley, W. B. Late results of the treatment of inoperable sarcoma by the mixed toxins of erysipelas and bacillus prodigiosus. Am J Med Sci. 131: 375-430, 1906
- [Background] Coley WB. The Treatment of Inoperable Sarcoma by Bacterial Toxins (the Mixed Toxins of the Streptococcus erysipelas and the Bacillus prodigiosus). Proc R Soc Med. 1910;3(Surg Sect):1-48. doi: 10.1177/003591571000301601. No abstract available. PMID 19974799
- [Background] Han RF, Pan JG. Can intravesical bacillus Calmette-Guerin reduce recurrence in patients with superficial bladder cancer? A meta-analysis of randomized trials. Urology. 2006 Jun;67(6):1216-23. doi: 10.1016/j.urology.2005.12.014. PMID 16765182
- [Background] Janeway CA Jr. The immune system evolved to discriminate infectious nonself from noninfectious self. Immunol Today. 1992 Jan;13(1):11-6. doi: 10.1016/0167-5699(92)90198-G. PMID 1739426
- [Background] Matzinger P. Friendly and dangerous signals: is the tissue in control? Nat Immunol. 2007 Jan;8(1):11-3. doi: 10.1038/ni0107-11. PMID 17179963
- [Background] Hammerich L, Binder A, Brody JD. In situ vaccination: Cancer immunotherapy both personalized and off-the-shelf. Mol Oncol. 2015 Dec;9(10):1966-81. doi: 10.1016/j.molonc.2015.10.016. Epub 2015 Nov 10. PMID 26632446
- [Background] Marabelle A, Kohrt H, Caux C, Levy R. Intratumoral immunization: a new paradigm for cancer therapy. Clin Cancer Res. 2014 Apr 1;20(7):1747-56. doi: 10.1158/1078-0432.CCR-13-2116. PMID 24691639
- [Background] Kaminski JM, Shinohara E, Summers JB, Niermann KJ, Morimoto A, Brousal J. The controversial abscopal effect. Cancer Treat Rev. 2005 May;31(3):159-72. doi: 10.1016/j.ctrv.2005.03.004. PMID 15923088
- [Background] Steinman RM. Decisions about dendritic cells: past, present, and future. Annu Rev Immunol. 2012;30:1-22. doi: 10.1146/annurev-immunol-100311-102839. Epub 2011 Nov 17. PMID 22136168
- [Background] Joffre OP, Segura E, Savina A, Amigorena S. Cross-presentation by dendritic cells. Nat Rev Immunol. 2012 Jul 13;12(8):557-69. doi: 10.1038/nri3254. PMID 22790179
- [Background] Inaba K, Turley S, Yamaide F, Iyoda T, Mahnke K, Inaba M, Pack M, Subklewe M, Sauter B, Sheff D, Albert M, Bhardwaj N, Mellman I, Steinman RM. Efficient presentation of phagocytosed cellular fragments on the major histocompatibility complex class II products of dendritic cells. J Exp Med. 1998 Dec 7;188(11):2163-73. doi: 10.1084/jem.188.11.2163. PMID 9841929
- [Background] Broz ML, Binnewies M, Boldajipour B, Nelson AE, Pollack JL, Erle DJ, Barczak A, Rosenblum MD, Daud A, Barber DL, Amigorena S, Van't Veer LJ, Sperling AI, Wolf DM, Krummel MF. Dissecting the tumor myeloid compartment reveals rare activating antigen-presenting cells critical for T cell immunity. Cancer Cell. 2014 Nov 10;26(5):638-52. doi: 10.1016/j.ccell.2014.09.007. Epub 2014 Oct 16. PMID 25446897
- [Background] Hildner K, Edelson BT, Purtha WE, Diamond M, Matsushita H, Kohyama M, Calderon B, Schraml BU, Unanue ER, Diamond MS, Schreiber RD, Murphy TL, Murphy KM. Batf3 deficiency reveals a critical role for CD8alpha+ dendritic cells in cytotoxic T cell immunity. Science. 2008 Nov 14;322(5904):1097-100. doi: 10.1126/science.1164206. PMID 19008445
- [Background] Schraml BU, Reis e Sousa C. Defining dendritic cells. Curr Opin Immunol. 2015 Feb;32:13-20. doi: 10.1016/j.coi.2014.11.001. Epub 2014 Dec 3. PMID 25553392
- [Background] Poulin LF, Salio M, Griessinger E, Anjos-Afonso F, Craciun L, Chen JL, Keller AM, Joffre O, Zelenay S, Nye E, Le Moine A, Faure F, Donckier V, Sancho D, Cerundolo V, Bonnet D, Reis e Sousa C. Characterization of human DNGR-1+ BDCA3+ leukocytes as putative equivalents of mouse CD8alpha+ dendritic cells. J Exp Med. 2010 Jun 7;207(6):1261-71. doi: 10.1084/jem.20092618. Epub 2010 May 17. PMID 20479117
- [Background] Jongbloed SL, Kassianos AJ, McDonald KJ, Clark GJ, Ju X, Angel CE, Chen CJ, Dunbar PR, Wadley RB, Jeet V, Vulink AJ, Hart DN, Radford KJ. Human CD141+ (BDCA-3)+ dendritic cells (DCs) represent a unique myeloid DC subset that cross-presents necrotic cell antigens. J Exp Med. 2010 Jun 7;207(6):1247-60. doi: 10.1084/jem.20092140. Epub 2010 May 17. PMID 20479116
- [Background] Zitvogel L, Kroemer G. CD103+ dendritic cells producing interleukin-12 in anticancer immunosurveillance. Cancer Cell. 2014 Nov 10;26(5):591-3. doi: 10.1016/j.ccell.2014.10.008. Epub 2014 Nov 10. PMID 25517740
- [Background] Martinez-Lopez M, Iborra S, Conde-Garrosa R, Sancho D. Batf3-dependent CD103+ dendritic cells are major producers of IL-12 that drive local Th1 immunity against Leishmania major infection in mice. Eur J Immunol. 2015 Jan;45(1):119-29. doi: 10.1002/eji.201444651. Epub 2014 Nov 28. PMID 25312824
- [Background] Ghiringhelli F, Puig PE, Roux S, Parcellier A, Schmitt E, Solary E, Kroemer G, Martin F, Chauffert B, Zitvogel L. Tumor cells convert immature myeloid dendritic cells into TGF-beta-secreting cells inducing CD4+CD25+ regulatory T cell proliferation. J Exp Med. 2005 Oct 3;202(7):919-29. doi: 10.1084/jem.20050463. Epub 2005 Sep 26. PMID 16186184
- [Background] Herber DL, Cao W, Nefedova Y, Novitskiy SV, Nagaraj S, Tyurin VA, Corzo A, Cho HI, Celis E, Lennox B, Knight SC, Padhya T, McCaffrey TV, McCaffrey JC, Antonia S, Fishman M, Ferris RL, Kagan VE, Gabrilovich DI. Lipid accumulation and dendritic cell dysfunction in cancer. Nat Med. 2010 Aug;16(8):880-6. doi: 10.1038/nm.2172. Epub 2010 Jul 11. PMID 20622859
- [Background] Diaz-Valdes N, Manterola L, Belsue V, Riezu-Boj JI, Larrea E, Echeverria I, Llopiz D, Lopez-Sagaseta J, Lerat H, Pawlotsky JM, Prieto J, Lasarte JJ, Borras-Cuesta F, Sarobe P. Improved dendritic cell-based immunization against hepatitis C virus using peptide inhibitors of interleukin 10. Hepatology. 2011 Jan;53(1):23-31. doi: 10.1002/hep.23980. Epub 2010 Dec 13. PMID 21154952
- [Background] Ruffell B, Chang-Strachan D, Chan V, Rosenbusch A, Ho CM, Pryer N, Daniel D, Hwang ES, Rugo HS, Coussens LM. Macrophage IL-10 blocks CD8+ T cell-dependent responses to chemotherapy by suppressing IL-12 expression in intratumoral dendritic cells. Cancer Cell. 2014 Nov 10;26(5):623-37. doi: 10.1016/j.ccell.2014.09.006. Epub 2014 Oct 16. PMID 25446896
- [Background] Salmon H, Idoyaga J, Rahman A, Leboeuf M, Remark R, Jordan S, Casanova-Acebes M, Khudoynazarova M, Agudo J, Tung N, Chakarov S, Rivera C, Hogstad B, Bosenberg M, Hashimoto D, Gnjatic S, Bhardwaj N, Palucka AK, Brown BD, Brody J, Ginhoux F, Merad M. Expansion and Activation of CD103(+) Dendritic Cell Progenitors at the Tumor Site Enhances Tumor Responses to Therapeutic PD-L1 and BRAF Inhibition. Immunity. 2016 Apr 19;44(4):924-38. doi: 10.1016/j.immuni.2016.03.012. PMID 27096321
- [Background] Sanchez-Paulete AR, Cueto FJ, Martinez-Lopez M, Labiano S, Morales-Kastresana A, Rodriguez-Ruiz ME, Jure-Kunkel M, Azpilikueta A, Aznar MA, Quetglas JI, Sancho D, Melero I. Cancer Immunotherapy with Immunomodulatory Anti-CD137 and Anti-PD-1 Monoclonal Antibodies Requires BATF3-Dependent Dendritic Cells. Cancer Discov. 2016 Jan;6(1):71-9. doi: 10.1158/2159-8290.CD-15-0510. Epub 2015 Oct 22. PMID 26493961
- [Background] Sistigu A, Yamazaki T, Vacchelli E, Chaba K, Enot DP, Adam J, Vitale I, Goubar A, Baracco EE, Remedios C, Fend L, Hannani D, Aymeric L, Ma Y, Niso-Santano M, Kepp O, Schultze JL, Tuting T, Belardelli F, Bracci L, La Sorsa V, Ziccheddu G, Sestili P, Urbani F, Delorenzi M, Lacroix-Triki M, Quidville V, Conforti R, Spano JP, Pusztai L, Poirier-Colame V, Delaloge S, Penault-Llorca F, Ladoire S, Arnould L, Cyrta J, Dessoliers MC, Eggermont A, Bianchi ME, Pittet M, Engblom C, Pfirschke C, Preville X, Uze G, Schreiber RD, Chow MT, Smyth MJ, Proietti E, Andre F, Kroemer G, Zitvogel L. Cancer cell-autonomous contribution of type I interferon signaling to the efficacy of chemotherapy. Nat Med. 2014 Nov;20(11):1301-9. doi: 10.1038/nm.3708. Epub 2014 Oct 26. PMID 25344738
- [Background] Le Bon A, Etchart N, Rossmann C, Ashton M, Hou S, Gewert D, Borrow P, Tough DF. Cross-priming of CD8+ T cells stimulated by virus-induced type I interferon. Nat Immunol. 2003 Oct;4(10):1009-15. doi: 10.1038/ni978. Epub 2003 Sep 21. PMID 14502286
- [Background] Kroemer G, Galluzzi L, Kepp O, Zitvogel L. Immunogenic cell death in cancer therapy. Annu Rev Immunol. 2013;31:51-72. doi: 10.1146/annurev-immunol-032712-100008. Epub 2012 Nov 12. PMID 23157435
- [Background] Schiavoni G, Sistigu A, Valentini M, Mattei F, Sestili P, Spadaro F, Sanchez M, Lorenzi S, D'Urso MT, Belardelli F, Gabriele L, Proietti E, Bracci L. Cyclophosphamide synergizes with type I interferons through systemic dendritic cell reactivation and induction of immunogenic tumor apoptosis. Cancer Res. 2011 Feb 1;71(3):768-78. doi: 10.1158/0008-5472.CAN-10-2788. Epub 2010 Dec 13. PMID 21156650
- [Background] Kumar H, Kawai T, Akira S. Pathogen recognition by the innate immune system. Int Rev Immunol. 2011 Feb;30(1):16-34. doi: 10.3109/08830185.2010.529976. PMID 21235323
- [Background] Apetoh L, Ghiringhelli F, Tesniere A, Criollo A, Ortiz C, Lidereau R, Mariette C, Chaput N, Mira JP, Delaloge S, Andre F, Tursz T, Kroemer G, Zitvogel L. The interaction between HMGB1 and TLR4 dictates the outcome of anticancer chemotherapy and radiotherapy. Immunol Rev. 2007 Dec;220:47-59. doi: 10.1111/j.1600-065X.2007.00573.x. PMID 17979839
- [Background] Lasarte JJ, Casares N, Gorraiz M, Hervas-Stubbs S, Arribillaga L, Mansilla C, Durantez M, Llopiz D, Sarobe P, Borras-Cuesta F, Prieto J, Leclerc C. The extra domain A from fibronectin targets antigens to TLR4-expressing cells and induces cytotoxic T cell responses in vivo. J Immunol. 2007 Jan 15;178(2):748-56. doi: 10.4049/jimmunol.178.2.748. PMID 17202335
- [Background] Chicoine MR, Won EK, Zahner MC. Intratumoral injection of lipopolysaccharide causes regression of subcutaneously implanted mouse glioblastoma multiforme. Neurosurgery. 2001 Mar;48(3):607-14; discussion 614-5. doi: 10.1097/00006123-200103000-00032. PMID 11270552
- [Background] Van De Voort TJ, Felder MA, Yang RK, Sondel PM, Rakhmilevich AL. Intratumoral delivery of low doses of anti-CD40 mAb combined with monophosphoryl lipid a induces local and systemic antitumor effects in immunocompetent and T cell-deficient mice. J Immunother. 2013 Jan;36(1):29-40. doi: 10.1097/CJI.0b013e3182780f61. PMID 23211623
- [Background] Apetoh L, Ghiringhelli F, Tesniere A, Obeid M, Ortiz C, Criollo A, Mignot G, Maiuri MC, Ullrich E, Saulnier P, Yang H, Amigorena S, Ryffel B, Barrat FJ, Saftig P, Levi F, Lidereau R, Nogues C, Mira JP, Chompret A, Joulin V, Clavel-Chapelon F, Bourhis J, Andre F, Delaloge S, Tursz T, Kroemer G, Zitvogel L. Toll-like receptor 4-dependent contribution of the immune system to anticancer chemotherapy and radiotherapy. Nat Med. 2007 Sep;13(9):1050-9. doi: 10.1038/nm1622. Epub 2007 Aug 19. PMID 17704786
- [Background] Weide B, Eigentler TK, Pflugfelder A, Zelba H, Martens A, Pawelec G, Giovannoni L, Ruffini PA, Elia G, Neri D, Gutzmer R, Becker JC, Garbe C. Intralesional treatment of stage III metastatic melanoma patients with L19-IL2 results in sustained clinical and systemic immunologic responses. Cancer Immunol Res. 2014 Jul;2(7):668-78. doi: 10.1158/2326-6066.CIR-13-0206. Epub 2014 Apr 4. PMID 24906352
- [Background] Bauer S, Kirschning CJ, Hacker H, Redecke V, Hausmann S, Akira S, Wagner H, Lipford GB. Human TLR9 confers responsiveness to bacterial DNA via species-specific CpG motif recognition. Proc Natl Acad Sci U S A. 2001 Jul 31;98(16):9237-42. doi: 10.1073/pnas.161293498. Epub 2001 Jul 24. PMID 11470918
- [Background] Houot R, Levy R. T-cell modulation combined with intratumoral CpG cures lymphoma in a mouse model without the need for chemotherapy. Blood. 2009 Apr 9;113(15):3546-52. doi: 10.1182/blood-2008-07-170274. Epub 2008 Oct 21. PMID 18941113
- [Background] Li J, Song W, Czerwinski DK, Varghese B, Uematsu S, Akira S, Krieg AM, Levy R. Lymphoma immunotherapy with CpG oligodeoxynucleotides requires TLR9 either in the host or in the tumor itself. J Immunol. 2007 Aug 15;179(4):2493-500. doi: 10.4049/jimmunol.179.4.2493. PMID 17675511
- [Background] Meng Y, Carpentier AF, Chen L, Boisserie G, Simon JM, Mazeron JJ, Delattre JY. Successful combination of local CpG-ODN and radiotherapy in malignant glioma. Int J Cancer. 2005 Oct 10;116(6):992-7. doi: 10.1002/ijc.21131. PMID 15856470
- [Background] Brody JD, Ai WZ, Czerwinski DK, Torchia JA, Levy M, Advani RH, Kim YH, Hoppe RT, Knox SJ, Shin LK, Wapnir I, Tibshirani RJ, Levy R. In situ vaccination with a TLR9 agonist induces systemic lymphoma regression: a phase I/II study. J Clin Oncol. 2010 Oct 1;28(28):4324-32. doi: 10.1200/JCO.2010.28.9793. Epub 2010 Aug 9. PMID 20697067
- [Background] Daud AI, DeConti RC, Andrews S, Urbas P, Riker AI, Sondak VK, Munster PN, Sullivan DM, Ugen KE, Messina JL, Heller R. Phase I trial of interleukin-12 plasmid electroporation in patients with metastatic melanoma. J Clin Oncol. 2008 Dec 20;26(36):5896-903. doi: 10.1200/JCO.2007.15.6794. Epub 2008 Nov 24. PMID 19029422
- [Background] Rehwinkel J, Reis e Sousa C. RIGorous detection: exposing virus through RNA sensing. Science. 2010 Jan 15;327(5963):284-6. doi: 10.1126/science.1185068. PMID 20075242
- [Background] Alexopoulou L, Holt AC, Medzhitov R, Flavell RA. Recognition of double-stranded RNA and activation of NF-kappaB by Toll-like receptor 3. Nature. 2001 Oct 18;413(6857):732-8. doi: 10.1038/35099560. PMID 11607032
- [Background] Amos SM, Pegram HJ, Westwood JA, John LB, Devaud C, Clarke CJ, Restifo NP, Smyth MJ, Darcy PK, Kershaw MH. Adoptive immunotherapy combined with intratumoral TLR agonist delivery eradicates established melanoma in mice. Cancer Immunol Immunother. 2011 May;60(5):671-83. doi: 10.1007/s00262-011-0984-8. Epub 2011 Feb 16. PMID 21327636
- [Background] Bald T, Landsberg J, Lopez-Ramos D, Renn M, Glodde N, Jansen P, Gaffal E, Steitz J, Tolba R, Kalinke U, Limmer A, Jonsson G, Holzel M, Tuting T. Immune cell-poor melanomas benefit from PD-1 blockade after targeted type I IFN activation. Cancer Discov. 2014 Jun;4(6):674-87. doi: 10.1158/2159-8290.CD-13-0458. Epub 2014 Mar 3. PMID 24589924
- [Background] Salazar AM, Erlich RB, Mark A, Bhardwaj N, Herberman RB. Therapeutic in situ autovaccination against solid cancers with intratumoral poly-ICLC: case report, hypothesis, and clinical trial. Cancer Immunol Res. 2014 Aug;2(8):720-4. doi: 10.1158/2326-6066.CIR-14-0024. Epub 2014 May 6. PMID 24801836
- [Background] Tormo D, Checinska A, Alonso-Curbelo D, Perez-Guijarro E, Canon E, Riveiro-Falkenbach E, Calvo TG, Larribere L, Megias D, Mulero F, Piris MA, Dash R, Barral PM, Rodriguez-Peralto JL, Ortiz-Romero P, Tuting T, Fisher PB, Soengas MS. Targeted activation of innate immunity for therapeutic induction of autophagy and apoptosis in melanoma cells. Cancer Cell. 2009 Aug 4;16(2):103-14. doi: 10.1016/j.ccr.2009.07.004. PMID 19647221
- [Background] Jelinek I, Leonard JN, Price GE, Brown KN, Meyer-Manlapat A, Goldsmith PK, Wang Y, Venzon D, Epstein SL, Segal DM. TLR3-specific double-stranded RNA oligonucleotide adjuvants induce dendritic cell cross-presentation, CTL responses, and antiviral protection. J Immunol. 2011 Feb 15;186(4):2422-9. doi: 10.4049/jimmunol.1002845. Epub 2011 Jan 17. PMID 21242525
- [Background] Sidky YA, Borden EC, Weeks CE, Reiter MJ, Hatcher JF, Bryan GT. Inhibition of murine tumor growth by an interferon-inducing imidazoquinolinamine. Cancer Res. 1992 Jul 1;52(13):3528-33. PMID 1377595
- [Background] Ahonen CL, Gibson SJ, Smith RM, Pederson LK, Lindh JM, Tomai MA, Vasilakos JP. Dendritic cell maturation and subsequent enhanced T-cell stimulation induced with the novel synthetic immune response modifier R-848. Cell Immunol. 1999 Oct 10;197(1):62-72. doi: 10.1006/cimm.1999.1555. PMID 10555997
- [Background] Smyth EC, Flavin M, Pulitzer MP, Gardner GJ, Costantino PD, Chi DS, Bogatch K, Chapman PB, Wolchok JD, Schwartz GK, Carvajal RD. Treatment of locally recurrent mucosal melanoma with topical imiquimod. J Clin Oncol. 2011 Nov 20;29(33):e809-11. doi: 10.1200/JCO.2011.36.8829. Epub 2011 Oct 17. No abstract available. PMID 22010009
- [Background] Redondo P, del Olmo J, Lopez-Diaz de Cerio A, Inoges S, Marquina M, Melero I, Bendandi M. Imiquimod enhances the systemic immunity attained by local cryosurgery destruction of melanoma lesions. J Invest Dermatol. 2007 Jul;127(7):1673-80. doi: 10.1038/sj.jid.5700777. Epub 2007 Mar 22. PMID 17380112
- [Background] Dewan MZ, Vanpouille-Box C, Kawashima N, DiNapoli S, Babb JS, Formenti SC, Adams S, Demaria S. Synergy of topical toll-like receptor 7 agonist with radiation and low-dose cyclophosphamide in a mouse model of cutaneous breast cancer. Clin Cancer Res. 2012 Dec 15;18(24):6668-78. doi: 10.1158/1078-0432.CCR-12-0984. Epub 2012 Oct 9. PMID 23048078
- [Background] Adams S, Kozhaya L, Martiniuk F, Meng TC, Chiriboga L, Liebes L, Hochman T, Shuman N, Axelrod D, Speyer J, Novik Y, Tiersten A, Goldberg JD, Formenti SC, Bhardwaj N, Unutmaz D, Demaria S. Topical TLR7 agonist imiquimod can induce immune-mediated rejection of skin metastases in patients with breast cancer. Clin Cancer Res. 2012 Dec 15;18(24):6748-57. doi: 10.1158/1078-0432.CCR-12-1149. Epub 2012 Jul 5. PMID 22767669
- [Background] Corrales L, Glickman LH, McWhirter SM, Kanne DB, Sivick KE, Katibah GE, Woo SR, Lemmens E, Banda T, Leong JJ, Metchette K, Dubensky TW Jr, Gajewski TF. Direct Activation of STING in the Tumor Microenvironment Leads to Potent and Systemic Tumor Regression and Immunity. Cell Rep. 2015 May 19;11(7):1018-30. doi: 10.1016/j.celrep.2015.04.031. Epub 2015 May 7. PMID 25959818
- [Background] Ablasser A, Goldeck M, Cavlar T, Deimling T, Witte G, Rohl I, Hopfner KP, Ludwig J, Hornung V. cGAS produces a 2'-5'-linked cyclic dinucleotide second messenger that activates STING. Nature. 2013 Jun 20;498(7454):380-4. doi: 10.1038/nature12306. Epub 2013 May 30. PMID 23722158
- [Background] Zhang X, Shi H, Wu J, Zhang X, Sun L, Chen C, Chen ZJ. Cyclic GMP-AMP containing mixed phosphodiester linkages is an endogenous high-affinity ligand for STING. Mol Cell. 2013 Jul 25;51(2):226-35. doi: 10.1016/j.molcel.2013.05.022. Epub 2013 Jun 6. PMID 23747010
- [Background] Deng L, Liang H, Xu M, Yang X, Burnette B, Arina A, Li XD, Mauceri H, Beckett M, Darga T, Huang X, Gajewski TF, Chen ZJ, Fu YX, Weichselbaum RR. STING-Dependent Cytosolic DNA Sensing Promotes Radiation-Induced Type I Interferon-Dependent Antitumor Immunity in Immunogenic Tumors. Immunity. 2014 Nov 20;41(5):843-52. doi: 10.1016/j.immuni.2014.10.019. Epub 2014 Nov 6. PMID 25517616
- [Background] Woo SR, Fuertes MB, Corrales L, Spranger S, Furdyna MJ, Leung MY, Duggan R, Wang Y, Barber GN, Fitzgerald KA, Alegre ML, Gajewski TF. STING-dependent cytosolic DNA sensing mediates innate immune recognition of immunogenic tumors. Immunity. 2014 Nov 20;41(5):830-42. doi: 10.1016/j.immuni.2014.10.017. Epub 2014 Nov 5. PMID 25517615
- [Background] Lichty BD, Breitbach CJ, Stojdl DF, Bell JC. Going viral with cancer immunotherapy. Nat Rev Cancer. 2014 Aug;14(8):559-67. doi: 10.1038/nrc3770. Epub 2014 Jul 3. PMID 24990523
- [Background] Prestwich RJ, Harrington KJ, Pandha HS, Vile RG, Melcher AA, Errington F. Oncolytic viruses: a novel form of immunotherapy. Expert Rev Anticancer Ther. 2008 Oct;8(10):1581-8. doi: 10.1586/14737140.8.10.1581. PMID 18925850
- [Background] Smerdou C, Ochoa C, Quetglas JI, Fontanellas A, Gonzalez-Aseguinolaza G, Vile RG, Melero I. Immunology and gene therapy: shoulder to shoulder into the fray. Mol Ther. 2010 Mar;18(3):456-9. doi: 10.1038/mt.2010.7. No abstract available. PMID 20195262
- [Background] Goins WF, Huang S, Cohen JB, Glorioso JC. Engineering HSV-1 vectors for gene therapy. Methods Mol Biol. 2014;1144:63-79. doi: 10.1007/978-1-4939-0428-0_5. PMID 24671677
- [Background] Kim JH, Oh JY, Park BH, Lee DE, Kim JS, Park HE, Roh MS, Je JE, Yoon JH, Thorne SH, Kirn D, Hwang TH. Systemic armed oncolytic and immunologic therapy for cancer with JX-594, a targeted poxvirus expressing GM-CSF. Mol Ther. 2006 Sep;14(3):361-70. doi: 10.1016/j.ymthe.2006.05.008. PMID 16905462
- [Background] Rodriguez-Madoz JR, Prieto J, Smerdou C. Semliki forest virus vectors engineered to express higher IL-12 levels induce efficient elimination of murine colon adenocarcinomas. Mol Ther. 2005 Jul;12(1):153-63. doi: 10.1016/j.ymthe.2005.02.011. PMID 15963931
- [Background] Sangro B, Mazzolini G, Ruiz J, Herraiz M, Quiroga J, Herrero I, Benito A, Larrache J, Pueyo J, Subtil JC, Olague C, Sola J, Sadaba B, Lacasa C, Melero I, Qian C, Prieto J. Phase I trial of intratumoral injection of an adenovirus encoding interleukin-12 for advanced digestive tumors. J Clin Oncol. 2004 Apr 15;22(8):1389-97. doi: 10.1200/JCO.2004.04.059. PMID 15084613
- [Background] Agrawal N, Bettegowda C, Cheong I, Geschwind JF, Drake CG, Hipkiss EL, Tatsumi M, Dang LH, Diaz LA Jr, Pomper M, Abusedera M, Wahl RL, Kinzler KW, Zhou S, Huso DL, Vogelstein B. Bacteriolytic therapy can generate a potent immune response against experimental tumors. Proc Natl Acad Sci U S A. 2004 Oct 19;101(42):15172-7. doi: 10.1073/pnas.0406242101. Epub 2004 Oct 7. PMID 15471990
- [Background] Barajas M, Mazzolini G, Genove G, Bilbao R, Narvaiza I, Schmitz V, Sangro B, Melero I, Qian C, Prieto J. Gene therapy of orthotopic hepatocellular carcinoma in rats using adenovirus coding for interleukin 12. Hepatology. 2001 Jan;33(1):52-61. doi: 10.1053/jhep.2001.20796. PMID 11124820
- [Background] Quetglas JI, Ruiz-Guillen M, Aranda A, Casales E, Bezunartea J, Smerdou C. Alphavirus vectors for cancer therapy. Virus Res. 2010 Nov;153(2):179-96. doi: 10.1016/j.virusres.2010.07.027. Epub 2010 Aug 6. PMID 20692305
- [Background] Ott PA, Hodi FS. Talimogene Laherparepvec for the Treatment of Advanced Melanoma. Clin Cancer Res. 2016 Jul 1;22(13):3127-31. doi: 10.1158/1078-0432.CCR-15-2709. Epub 2016 May 4. PMID 27146699
- [Background] Lorence RM, Reichard KW, Katubig BB, Reyes HM, Phuangsab A, Mitchell BR, Cascino CJ, Walter RJ, Peeples ME. Complete regression of human neuroblastoma xenografts in athymic mice after local Newcastle disease virus therapy. J Natl Cancer Inst. 1994 Aug 17;86(16):1228-33. doi: 10.1093/jnci/86.16.1228. PMID 8040891
- [Background] Nistal-Villan E, Bunuales M, Poutou J, Gonzalez-Aparicio M, Bravo-Perez C, Quetglas JI, Carte B, Gonzalez-Aseguinolaza G, Prieto J, Larrea E, Hernandez-Alcoceba R. Enhanced therapeutic effect using sequential administration of antigenically distinct oncolytic viruses expressing oncostatin M in a Syrian hamster orthotopic pancreatic cancer model. Mol Cancer. 2015 Dec 16;14:210. doi: 10.1186/s12943-015-0479-x. PMID 26671477
- [Background] Zamarin D, Holmgaard RB, Subudhi SK, Park JS, Mansour M, Palese P, Merghoub T, Wolchok JD, Allison JP. Localized oncolytic virotherapy overcomes systemic tumor resistance to immune checkpoint blockade immunotherapy. Sci Transl Med. 2014 Mar 5;6(226):226ra32. doi: 10.1126/scitranslmed.3008095. PMID 24598590
- [Background] Lundstrom K. Alphaviruses in gene therapy. Viruses. 2009 Jun;1(1):13-25. doi: 10.3390/v1010013. Epub 2009 Apr 21. PMID 21994535
- [Background] Melero I, Quetglas JI, Reboredo M, Dubrot J, Rodriguez-Madoz JR, Mancheno U, Casales E, Riezu-Boj JI, Ruiz-Guillen M, Ochoa MC, Sanmamed MF, Thieblemont N, Smerdou C, Hervas-Stubbs S. Strict requirement for vector-induced type I interferon in efficacious antitumor responses to virally encoded IL12. Cancer Res. 2015 Feb 1;75(3):497-507. doi: 10.1158/0008-5472.CAN-13-3356. Epub 2014 Dec 19. PMID 25527611
- [Background] Andtbacka RH, Kaufman HL, Collichio F, Amatruda T, Senzer N, Chesney J, Delman KA, Spitler LE, Puzanov I, Agarwala SS, Milhem M, Cranmer L, Curti B, Lewis K, Ross M, Guthrie T, Linette GP, Daniels GA, Harrington K, Middleton MR, Miller WH Jr, Zager JS, Ye Y, Yao B, Li A, Doleman S, VanderWalde A, Gansert J, Coffin RS. Talimogene Laherparepvec Improves Durable Response Rate in Patients With Advanced Melanoma. J Clin Oncol. 2015 Sep 1;33(25):2780-8. doi: 10.1200/JCO.2014.58.3377. Epub 2015 May 26. PMID 26014293
- [Background] Narvaiza I, Mazzolini G, Barajas M, Duarte M, Zaratiegui M, Qian C, Melero I, Prieto J. Intratumoral coinjection of two adenoviruses, one encoding the chemokine IFN-gamma-inducible protein-10 and another encoding IL-12, results in marked antitumoral synergy. J Immunol. 2000 Mar 15;164(6):3112-22. doi: 10.4049/jimmunol.164.6.3112. PMID 10706701
- [Background] Park BH, Hwang T, Liu TC, Sze DY, Kim JS, Kwon HC, Oh SY, Han SY, Yoon JH, Hong SH, Moon A, Speth K, Park C, Ahn YJ, Daneshmand M, Rhee BG, Pinedo HM, Bell JC, Kirn DH. Use of a targeted oncolytic poxvirus, JX-594, in patients with refractory primary or metastatic liver cancer: a phase I trial. Lancet Oncol. 2008 Jun;9(6):533-42. doi: 10.1016/S1470-2045(08)70107-4. Epub 2008 May 19. PMID 18495536
- [Background] Quetglas JI, Labiano S, Aznar MA, Bolanos E, Azpilikueta A, Rodriguez I, Casales E, Sanchez-Paulete AR, Segura V, Smerdou C, Melero I. Virotherapy with a Semliki Forest Virus-Based Vector Encoding IL12 Synergizes with PD-1/PD-L1 Blockade. Cancer Immunol Res. 2015 May;3(5):449-54. doi: 10.1158/2326-6066.CIR-14-0216. Epub 2015 Feb 17. PMID 25691326
- [Background] Quetglas JI, Dubrot J, Bezunartea J, Sanmamed MF, Hervas-Stubbs S, Smerdou C, Melero I. Immunotherapeutic synergy between anti-CD137 mAb and intratumoral administration of a cytopathic Semliki Forest virus encoding IL-12. Mol Ther. 2012 Sep;20(9):1664-1675. doi: 10.1038/mt.2012.56. Epub 2012 Jun 26. PMID 22735380
- [Background] John LB, Howland LJ, Flynn JK, West AC, Devaud C, Duong CP, Stewart TJ, Westwood JA, Guo ZS, Bartlett DL, Smyth MJ, Kershaw MH, Darcy PK. Oncolytic virus and anti-4-1BB combination therapy elicits strong antitumor immunity against established cancer. Cancer Res. 2012 Apr 1;72(7):1651-60. doi: 10.1158/0008-5472.CAN-11-2788. Epub 2012 Feb 7. PMID 22315352
- [Background] Puzanov I, Milhem MM, Minor D, Hamid O, Li A, Chen L, Chastain M, Gorski KS, Anderson A, Chou J, Kaufman HL, Andtbacka RH. Talimogene Laherparepvec in Combination With Ipilimumab in Previously Untreated, Unresectable Stage IIIB-IV Melanoma. J Clin Oncol. 2016 Aug 1;34(22):2619-26. doi: 10.1200/JCO.2016.67.1529. Epub 2016 Jun 13. PMID 27298410
- [Background] Breitbach CJ, Moon A, Burke J, Hwang TH, Kirn DH. A Phase 2, Open-Label, Randomized Study of Pexa-Vec (JX-594) Administered by Intratumoral Injection in Patients with Unresectable Primary Hepatocellular Carcinoma. Methods Mol Biol. 2015;1317:343-57. doi: 10.1007/978-1-4939-2727-2_19. PMID 26072416
- [Background] Cripe TP, Ngo MC, Geller JI, Louis CU, Currier MA, Racadio JM, Towbin AJ, Rooney CM, Pelusio A, Moon A, Hwang TH, Burke JM, Bell JC, Kirn DH, Breitbach CJ. Phase 1 study of intratumoral Pexa-Vec (JX-594), an oncolytic and immunotherapeutic vaccinia virus, in pediatric cancer patients. Mol Ther. 2015 Mar;23(3):602-8. doi: 10.1038/mt.2014.243. Epub 2014 Dec 22. PMID 25531693
- [Background] Huang PI, Chang JF, Kirn DH, Liu TC. Targeted genetic and viral therapy for advanced head and neck cancers. Drug Discov Today. 2009 Jun;14(11-12):570-8. doi: 10.1016/j.drudis.2009.03.008. Epub 2009 Mar 17. PMID 19508919
- [Background] Liu TC, Thorne SH, Kirn DH. Oncolytic adenoviruses for cancer gene therapy. Methods Mol Biol. 2008;433:243-58. doi: 10.1007/978-1-59745-237-3_15. PMID 18679628
- [Background] Huarte E, Larrea E, Hernandez-Alcoceba R, Alfaro C, Murillo O, Arina A, Tirapu I, Azpilicueta A, Hervas-Stubbs S, Bortolanza S, Perez-Gracia JL, Civeira MP, Prieto J, Riezu-Boj JI, Melero I. Recombinant adenoviral vectors turn on the type I interferon system without inhibition of transgene expression and viral replication. Mol Ther. 2006 Jul;14(1):129-38. doi: 10.1016/j.ymthe.2006.02.015. Epub 2006 Apr 19. PMID 16627004
- [Background] Kawai T, Akira S. Toll-like receptors and their crosstalk with other innate receptors in infection and immunity. Immunity. 2011 May 27;34(5):637-50. doi: 10.1016/j.immuni.2011.05.006. PMID 21616434
- [Background] Takeuchi O, Akira S. MDA5/RIG-I and virus recognition. Curr Opin Immunol. 2008 Feb;20(1):17-22. doi: 10.1016/j.coi.2008.01.002. Epub 2008 Feb 12. PMID 18272355
- [Background] Sharma P, Allison JP. The future of immune checkpoint therapy. Science. 2015 Apr 3;348(6230):56-61. doi: 10.1126/science.aaa8172. PMID 25838373
- [Background] Topalian SL, Drake CG, Pardoll DM. Immune checkpoint blockade: a common denominator approach to cancer therapy. Cancer Cell. 2015 Apr 13;27(4):450-61. doi: 10.1016/j.ccell.2015.03.001. Epub 2015 Apr 6. PMID 25858804
- [Background] Kohrt HE, Tumeh PC, Benson D, Bhardwaj N, Brody J, Formenti S, Fox BA, Galon J, June CH, Kalos M, Kirsch I, Kleen T, Kroemer G, Lanier L, Levy R, Lyerly HK, Maecker H, Marabelle A, Melenhorst J, Miller J, Melero I, Odunsi K, Palucka K, Peoples G, Ribas A, Robins H, Robinson W, Serafini T, Sondel P, Vivier E, Weber J, Wolchok J, Zitvogel L, Disis ML, Cheever MA; Cancer Immunotherapy Trials Network (CITN). Immunodynamics: a cancer immunotherapy trials network review of immune monitoring in immuno-oncology clinical trials. J Immunother Cancer. 2016 Mar 15;4:15. doi: 10.1186/s40425-016-0118-0. eCollection 2016. PMID 26981245
- [Background] Melief CJ. Selective activation of oxygen-deprived tumor-infiltrating lymphocytes through local intratumoral delivery of CD137 monoclonal antibodies. Cancer Discov. 2012 Jul;2(7):586-7. doi: 10.1158/2159-8290.CD-12-0229. PMID 22787088
- [Background] Fransen MF, van der Sluis TC, Ossendorp F, Arens R, Melief CJ. Controlled local delivery of CTLA-4 blocking antibody induces CD8+ T-cell-dependent tumor eradication and decreases risk of toxic side effects. Clin Cancer Res. 2013 Oct 1;19(19):5381-9. doi: 10.1158/1078-0432.CCR-12-0781. Epub 2013 Jun 20. PMID 23788581
- [Background] Fransen MF, Sluijter M, Morreau H, Arens R, Melief CJ. Local activation of CD8 T cells and systemic tumor eradication without toxicity via slow release and local delivery of agonistic CD40 antibody. Clin Cancer Res. 2011 Apr 15;17(8):2270-80. doi: 10.1158/1078-0432.CCR-10-2888. Epub 2011 Mar 9. PMID 21389097
- [Background] Fransen MF, Cordfunke RA, Sluijter M, van Steenbergen MJ, Drijfhout JW, Ossendorp F, Hennink WE, Melief CJ. Effectiveness of slow-release systems in CD40 agonistic antibody immunotherapy of cancer. Vaccine. 2014 Mar 26;32(15):1654-60. doi: 10.1016/j.vaccine.2014.01.056. Epub 2014 Feb 7. PMID 24508038
- [Background] Marabelle A, Kohrt H, Levy R. New insights into the mechanism of action of immune checkpoint antibodies. Oncoimmunology. 2014 Aug 3;3(8):e954869. doi: 10.4161/21624011.2014.954869. eCollection 2014. PMID 25610751
- [Background] Marabelle A, Kohrt H, Sagiv-Barfi I, Ajami B, Axtell RC, Zhou G, Rajapaksa R, Green MR, Torchia J, Brody J, Luong R, Rosenblum MD, Steinman L, Levitsky HI, Tse V, Levy R. Depleting tumor-specific Tregs at a single site eradicates disseminated tumors. J Clin Invest. 2013 Jun;123(6):2447-63. doi: 10.1172/JCI64859. PMID 23728179
- [Background] Lehmann S, Perera R, Grimm HP, Sam J, Colombetti S, Fauti T, Fahrni L, Schaller T, Freimoser-Grundschober A, Zielonka J, Stoma S, Rudin M, Klein C, Umana P, Gerdes C, Bacac M. In Vivo Fluorescence Imaging of the Activity of CEA TCB, a Novel T-Cell Bispecific Antibody, Reveals Highly Specific Tumor Targeting and Fast Induction of T-Cell-Mediated Tumor Killing. Clin Cancer Res. 2016 Sep 1;22(17):4417-27. doi: 10.1158/1078-0432.CCR-15-2622. Epub 2016 Apr 26. PMID 27117182
- [Background] Palazon A, Martinez-Forero I, Teijeira A, Morales-Kastresana A, Alfaro C, Sanmamed MF, Perez-Gracia JL, Penuelas I, Hervas-Stubbs S, Rouzaut A, de Landazuri MO, Jure-Kunkel M, Aragones J, Melero I. The HIF-1alpha hypoxia response in tumor-infiltrating T lymphocytes induces functional CD137 (4-1BB) for immunotherapy. Cancer Discov. 2012 Jul;2(7):608-23. doi: 10.1158/2159-8290.CD-11-0314. Epub 2012 Jun 19. PMID 22719018
- [Background] Beatty GL, Torigian DA, Chiorean EG, Saboury B, Brothers A, Alavi A, Troxel AB, Sun W, Teitelbaum UR, Vonderheide RH, O'Dwyer PJ. A phase I study of an agonist CD40 monoclonal antibody (CP-870,893) in combination with gemcitabine in patients with advanced pancreatic ductal adenocarcinoma. Clin Cancer Res. 2013 Nov 15;19(22):6286-95. doi: 10.1158/1078-0432.CCR-13-1320. Epub 2013 Aug 27. PMID 23983255
- [Background] Dubrot J, Milheiro F, Alfaro C, Palazon A, Martinez-Forero I, Perez-Gracia JL, Morales-Kastresana A, Romero-Trevejo JL, Ochoa MC, Hervas-Stubbs S, Prieto J, Jure-Kunkel M, Chen L, Melero I. Treatment with anti-CD137 mAbs causes intense accumulations of liver T cells without selective antitumor immunotherapeutic effects in this organ. Cancer Immunol Immunother. 2010 Aug;59(8):1223-33. doi: 10.1007/s00262-010-0846-9. Epub 2010 Mar 25. PMID 20336294
- [Background] Nowak AK, Cook AM, McDonnell AM, Millward MJ, Creaney J, Francis RJ, Hasani A, Segal A, Musk AW, Turlach BA, McCoy MJ, Robinson BW, Lake RA. A phase 1b clinical trial of the CD40-activating antibody CP-870,893 in combination with cisplatin and pemetrexed in malignant pleural mesothelioma. Ann Oncol. 2015 Dec;26(12):2483-90. doi: 10.1093/annonc/mdv387. Epub 2015 Sep 18. PMID 26386124
- [Background] Vonderheide RH, Flaherty KT, Khalil M, Stumacher MS, Bajor DL, Hutnick NA, Sullivan P, Mahany JJ, Gallagher M, Kramer A, Green SJ, O'Dwyer PJ, Running KL, Huhn RD, Antonia SJ. Clinical activity and immune modulation in cancer patients treated with CP-870,893, a novel CD40 agonist monoclonal antibody. J Clin Oncol. 2007 Mar 1;25(7):876-83. doi: 10.1200/JCO.2006.08.3311. PMID 17327609
- [Background] Bol KF, Schreibelt G, Gerritsen WR, de Vries IJ, Figdor CG. Dendritic Cell-Based Immunotherapy: State of the Art and Beyond. Clin Cancer Res. 2016 Apr 15;22(8):1897-906. doi: 10.1158/1078-0432.CCR-15-1399. PMID 27084743
- [Background] Alfaro C, Perez-Gracia JL, Suarez N, Rodriguez J, Fernandez de Sanmamed M, Sangro B, Martin-Algarra S, Calvo A, Redrado M, Agliano A, Gonzalez A, Rodriguez I, Bolanos E, Hervas-Stubbs S, Perez-Calvo J, Benito A, Penuelas I, Vigil C, Richter J, Martinez-Forero I, Melero I. Pilot clinical trial of type 1 dendritic cells loaded with autologous tumor lysates combined with GM-CSF, pegylated IFN, and cyclophosphamide for metastatic cancer patients. J Immunol. 2011 Dec 1;187(11):6130-42. doi: 10.4049/jimmunol.1102209. Epub 2011 Nov 2. PMID 22048768
- [Background] Bedrosian I, Mick R, Xu S, Nisenbaum H, Faries M, Zhang P, Cohen PA, Koski G, Czerniecki BJ. Intranodal administration of peptide-pulsed mature dendritic cell vaccines results in superior CD8+ T-cell function in melanoma patients. J Clin Oncol. 2003 Oct 15;21(20):3826-35. doi: 10.1200/JCO.2003.04.042. PMID 14551301
- [Background] Gilliet M, Kleinhans M, Lantelme E, Schadendorf D, Burg G, Nestle FO. Intranodal injection of semimature monocyte-derived dendritic cells induces T helper type 1 responses to protein neoantigen. Blood. 2003 Jul 1;102(1):36-42. doi: 10.1182/blood-2002-07-2274. Epub 2003 Jan 30. PMID 12560234
- [Background] Melero I, Duarte M, Ruiz J, Sangro B, Galofre J, Mazzolini G, Bustos M, Qian C, Prieto J. Intratumoral injection of bone-marrow derived dendritic cells engineered to produce interleukin-12 induces complete regression of established murine transplantable colon adenocarcinomas. Gene Ther. 1999 Oct;6(10):1779-84. doi: 10.1038/sj.gt.3301010. PMID 10516729
- [Background] Nishioka Y, Hirao M, Robbins PD, Lotze MT, Tahara H. Induction of systemic and therapeutic antitumor immunity using intratumoral injection of dendritic cells genetically modified to express interleukin 12. Cancer Res. 1999 Aug 15;59(16):4035-41. PMID 10463604
- [Background] Van Lint S, Renmans D, Broos K, Goethals L, Maenhout S, Benteyn D, Goyvaerts C, Du Four S, Van der Jeught K, Bialkowski L, Flamand V, Heirman C, Thielemans K, Breckpot K. Intratumoral Delivery of TriMix mRNA Results in T-cell Activation by Cross-Presenting Dendritic Cells. Cancer Immunol Res. 2016 Feb;4(2):146-56. doi: 10.1158/2326-6066.CIR-15-0163. Epub 2015 Dec 11. PMID 26659303
- [Background] Mazzolini G, Alfaro C, Sangro B, Feijoo E, Ruiz J, Benito A, Tirapu I, Arina A, Sola J, Herraiz M, Lucena F, Olague C, Subtil J, Quiroga J, Herrero I, Sadaba B, Bendandi M, Qian C, Prieto J, Melero I. Intratumoral injection of dendritic cells engineered to secrete interleukin-12 by recombinant adenovirus in patients with metastatic gastrointestinal carcinomas. J Clin Oncol. 2005 Feb 10;23(5):999-1010. doi: 10.1200/JCO.2005.00.463. Epub 2004 Dec 14. PMID 15598979
- [Background] Alfaro C, Suarez N, Martinez-Forero I, Palazon A, Rouzaut A, Solano S, Feijoo E, Gurpide A, Bolanos E, Erro L, Dubrot J, Hervas-Stubbs S, Gonzalez A, Perez-Gracia JL, Melero I. Carcinoma-derived interleukin-8 disorients dendritic cell migration without impairing T-cell stimulation. PLoS One. 2011 Mar 14;6(3):e17922. doi: 10.1371/journal.pone.0017922. PMID 21423807
- [Background] Melero I, Arina A, Murillo O, Dubrot J, Alfaro C, Perez-Gracia JL, Bendandi M, Hervas-Stubbs S. Immunogenic cell death and cross-priming are reaching the clinical immunotherapy arena. Clin Cancer Res. 2006 Apr 15;12(8):2385-9. doi: 10.1158/1078-0432.CCR-06-0314. No abstract available. PMID 16638842
- [Background] Spranger S, Bao R, Gajewski TF. Melanoma-intrinsic beta-catenin signalling prevents anti-tumour immunity. Nature. 2015 Jul 9;523(7559):231-5. doi: 10.1038/nature14404. Epub 2015 May 11. PMID 25970248
- [Background] Melero I, Vile RG, Colombo MP. Feeding dendritic cells with tumor antigens: self-service buffet or a la carte? Gene Ther. 2000 Jul;7(14):1167-70. doi: 10.1038/sj.gt.3301234. PMID 10918484
- [Background] Chi KH, Liu SJ, Li CP, Kuo HP, Wang YS, Chao Y, Hsieh SL. Combination of conformal radiotherapy and intratumoral injection of adoptive dendritic cell immunotherapy in refractory hepatoma. J Immunother. 2005 Mar-Apr;28(2):129-35. doi: 10.1097/01.cji.0000154248.74383.5e. PMID 15725956
- [Background] Breton G, Lee J, Zhou YJ, Schreiber JJ, Keler T, Puhr S, Anandasabapathy N, Schlesinger S, Caskey M, Liu K, Nussenzweig MC. Circulating precursors of human CD1c+ and CD141+ dendritic cells. J Exp Med. 2015 Mar 9;212(3):401-13. doi: 10.1084/jem.20141441. Epub 2015 Feb 16. PMID 25687281
- [Background] Gorelik L, Flavell RA. Transforming growth factor-beta in T-cell biology. Nat Rev Immunol. 2002 Jan;2(1):46-53. doi: 10.1038/nri704. PMID 11905837
- [Background] Li MO, Wan YY, Sanjabi S, Robertson AK, Flavell RA. Transforming growth factor-beta regulation of immune responses. Annu Rev Immunol. 2006;24:99-146. doi: 10.1146/annurev.immunol.24.021605.090737. PMID 16551245
- [Background] Maus MV, June CH. Making Better Chimeric Antigen Receptors for Adoptive T-cell Therapy. Clin Cancer Res. 2016 Apr 15;22(8):1875-84. doi: 10.1158/1078-0432.CCR-15-1433. PMID 27084741
- [Background] Rosenberg SA, Restifo NP. Adoptive cell transfer as personalized immunotherapy for human cancer. Science. 2015 Apr 3;348(6230):62-8. doi: 10.1126/science.aaa4967. PMID 25838374
- [Background] Melero I, Rouzaut A, Motz GT, Coukos G. T-cell and NK-cell infiltration into solid tumors: a key limiting factor for efficacious cancer immunotherapy. Cancer Discov. 2014 May;4(5):522-6. doi: 10.1158/2159-8290.CD-13-0985. PMID 24795012
- [Background] Arina A, Murillo O, Hervas-Stubbs S, Azpilikueta A, Dubrot J, Tirapu I, Huarte E, Alfaro C, Perez-Gracia JL, Gonzalez-Aseguinolaza G, Sarobe P, Lasarte JJ, Jamieson A, Prieto J, Raulet DH, Melero I. The combined actions of NK and T lymphocytes are necessary to reject an EGFP+ mesenchymal tumor through mechanisms dependent on NKG2D and IFN gamma. Int J Cancer. 2007 Sep 15;121(6):1282-95. doi: 10.1002/ijc.22795. PMID 17520674
- [Background] Golden EB, Pellicciotta I, Demaria S, Barcellos-Hoff MH, Formenti SC. The convergence of radiation and immunogenic cell death signaling pathways. Front Oncol. 2012 Aug 7;2:88. doi: 10.3389/fonc.2012.00088. eCollection 2012. PMID 22891162
- [Background] Kepp, O., L. Senovilla, I. Vitale, E. Vacchelli, S. Adjemian, P. Agostinis, L. Apetoh, F. Aranda, V. Barnaba, N. Bloy, L. Bracci, K. Breckpot, D. Brough, A. Buque, M. G. Castro, M. Cirone, M. I. Colombo, I. Cremer, S. Demaria, L. Dini, A. G. Eliopoulos, A. Faggioni, S. C. Formenti, J. Fucikova, L. Gabriele, U. S. Gaipl, J. Galon, A. Garg, F. Ghiringhelli, N. A. Giese, Z. S. Guo, A. Hemminki, M. Herrmann, J. W. Hodge, S. Holdenrieder, J. Honeychurch, H. M. Hu, X. Huang, T. M. Illidge, K. Kono, M. Korbelik, D. V. Krysko, S. Loi, P. R. Lowenstein, E. Lugli, Y. Ma, F. Madeo, A. A. Manfredi, I. Martins, D. Mavilio, L. Menger, N. Merendino, M. Michaud, G. Mignot, K. L. Mossman, G. Multhoff, R. Oehler, F. Palombo, T. Panaretakis, J. Pol, E. Proietti, J. E. Ricci, C. Riganti, P. Rovere-Querini, A. Rubartelli, A. Sistigu, M. J. Smyth, J. Sonnemann, R. Spisek, J. Stagg, A. Q. Sukkurwala, E. Tartour, A. Thorburn, S. H. Thorne, P. Vandenabeele, F. Velotti, S. T. Workenhe, H. Yang, W. X. Zong, L. Zitvogel, G. Kroemer, and L. Galluzzi. 2014. Consensus guidelines for the detection of immunogenic cell death. Oncoimmunology 3: e955691
- [Background] Antoniades J, Brady LW, Lightfoot DA. Lymphangiographic demonstration of the abscopal effect in patients with malignant lymphomas. Int J Radiat Oncol Biol Phys. 1977 Jan-Feb;2(1-2):141-7. doi: 10.1016/0360-3016(77)90020-7. No abstract available. PMID 403163
- [Background] Deng L, Liang H, Burnette B, Beckett M, Darga T, Weichselbaum RR, Fu YX. Irradiation and anti-PD-L1 treatment synergistically promote antitumor immunity in mice. J Clin Invest. 2014 Feb;124(2):687-95. doi: 10.1172/JCI67313. Epub 2014 Jan 2. PMID 24382348
- [Background] Ruocco MG, Pilones KA, Kawashima N, Cammer M, Huang J, Babb JS, Liu M, Formenti SC, Dustin ML, Demaria S. Suppressing T cell motility induced by anti-CTLA-4 monotherapy improves antitumor effects. J Clin Invest. 2012 Oct;122(10):3718-30. doi: 10.1172/JCI61931. Epub 2012 Sep 4. PMID 22945631
- [Background] Twyman-Saint Victor C, Rech AJ, Maity A, Rengan R, Pauken KE, Stelekati E, Benci JL, Xu B, Dada H, Odorizzi PM, Herati RS, Mansfield KD, Patsch D, Amaravadi RK, Schuchter LM, Ishwaran H, Mick R, Pryma DA, Xu X, Feldman MD, Gangadhar TC, Hahn SM, Wherry EJ, Vonderheide RH, Minn AJ. Radiation and dual checkpoint blockade activate non-redundant immune mechanisms in cancer. Nature. 2015 Apr 16;520(7547):373-7. doi: 10.1038/nature14292. Epub 2015 Mar 9. PMID 25754329
- [Background] Postow MA, Callahan MK, Barker CA, Yamada Y, Yuan J, Kitano S, Mu Z, Rasalan T, Adamow M, Ritter E, Sedrak C, Jungbluth AA, Chua R, Yang AS, Roman RA, Rosner S, Benson B, Allison JP, Lesokhin AM, Gnjatic S, Wolchok JD. Immunologic correlates of the abscopal effect in a patient with melanoma. N Engl J Med. 2012 Mar 8;366(10):925-31. doi: 10.1056/NEJMoa1112824. PMID 22397654
- [Background] Shi L, Chen L, Wu C, Zhu Y, Xu B, Zheng X, Sun M, Wen W, Dai X, Yang M, Lv Q, Lu B, Jiang J. PD-1 Blockade Boosts Radiofrequency Ablation-Elicited Adaptive Immune Responses against Tumor. Clin Cancer Res. 2016 Mar 1;22(5):1173-1184. doi: 10.1158/1078-0432.CCR-15-1352. PMID 26933175
- [Background] Mozzillo N, Simeone E, Benedetto L, Curvietto M, Giannarelli D, Gentilcore G, Camerlingo R, Capone M, Madonna G, Festino L, Caraco C, Di Monta G, Marone U, Di Marzo M, Grimaldi AM, Mori S, Ciliberto G, Ascierto PA. Assessing a novel immuno-oncology-based combination therapy: Ipilimumab plus electrochemotherapy. Oncoimmunology. 2015 May 22;4(6):e1008842. doi: 10.1080/2162402X.2015.1008842. eCollection 2015 Jun. PMID 26155423
- [Background] Korangy, F., M. ElGindi, D. Pratt, D. Venzon, A. Duffy, O. Makarova-Rusher, S. Kerkar, D. Kleiner, B. Wood, and T. Greten. 2016. Tremelimimab activates CD4 and CD8+T cells in patients with hepatocellular carcinoma. Cancer immunology research 4
- [Background] Barker HE, Paget JT, Khan AA, Harrington KJ. The tumour microenvironment after radiotherapy: mechanisms of resistance and recurrence. Nat Rev Cancer. 2015 Jul;15(7):409-25. doi: 10.1038/nrc3958. PMID 26105538
- [Background] Sandoval F, Terme M, Nizard M, Badoual C, Bureau MF, Freyburger L, Clement O, Marcheteau E, Gey A, Fraisse G, Bouguin C, Merillon N, Dransart E, Tran T, Quintin-Colonna F, Autret G, Thiebaud M, Suleman M, Riffault S, Wu TC, Launay O, Danel C, Taieb J, Richardson J, Zitvogel L, Fridman WH, Johannes L, Tartour E. Mucosal imprinting of vaccine-induced CD8(+) T cells is crucial to inhibit the growth of mucosal tumors. Sci Transl Med. 2013 Feb 13;5(172):172ra20. doi: 10.1126/scitranslmed.3004888. PMID 23408053
- [Background] Mikhak Z, Strassner JP, Luster AD. Lung dendritic cells imprint T cell lung homing and promote lung immunity through the chemokine receptor CCR4. J Exp Med. 2013 Aug 26;210(9):1855-69. doi: 10.1084/jem.20130091. Epub 2013 Aug 19. PMID 23960189
- [Background] Kaufman HL, Amatruda T, Reid T, Gonzalez R, Glaspy J, Whitman E, Harrington K, Nemunaitis J, Zloza A, Wolf M, Senzer NN. Systemic versus local responses in melanoma patients treated with talimogene laherparepvec from a multi-institutional phase II study. J Immunother Cancer. 2016 Mar 15;4:12. doi: 10.1186/s40425-016-0116-2. eCollection 2016. PMID 26981242
- [Background] Melero I, Berman DM, Aznar MA, Korman AJ, Perez Gracia JL, Haanen J. Evolving synergistic combinations of targeted immunotherapies to combat cancer. Nat Rev Cancer. 2015 Aug;15(8):457-72. doi: 10.1038/nrc3973. PMID 26205340
- [Background] Whiteside TL, Demaria S, Rodriguez-Ruiz ME, Zarour HM, Melero I. Emerging Opportunities and Challenges in Cancer Immunotherapy. Clin Cancer Res. 2016 Apr 15;22(8):1845-55. doi: 10.1158/1078-0432.CCR-16-0049. PMID 27084738
- [Background] Berraondo P, Ochoa MC, Rodriguez-Ruiz ME, Minute L, Lasarte JJ, Melero I. Immunostimulatory Monoclonal Antibodies and Immunomodulation: Harvesting the Crop. Cancer Res. 2016 May 15;76(10):2863-7. doi: 10.1158/0008-5472.CAN-15-3279. Epub 2016 May 2. PMID 27308833
- [Derived] Sanmamed MF, de Andrea CE, Ruiz-Guillamon D, Rodriguez-Ruiz ME, Ortego I, Eguren-Santamaria I, Benito A, Lopez-Janeiro A, Gonzalez Gomariz J, Villalba-Esparza M, Molina A, Krasko A, Ponz-Sarvise M, Lopez-Picazo JM, Gomis G, Molero-Glez P, Alexandru R, Perez-Dominguez P, Rodriguez I, Sanchez-Gregorio S, Perez-Gracia JL, Melero I. Safety, feasibility and pharmacodynamic activity of intratumoral injections of the agonist anti-CD137 (4-1BB) mAb urelumab in combination with nivolumab. Clin Cancer Res. 2026 Jan 16. doi: 10.1158/1078-0432.CCR-25-2502. Online ahead of print. PMID 41543348